CLINICAL TRIAL: NCT01497145
Title: A Phase 2, Randomized, Open-Label, Parallel, Comparative, Dose-Response Study to Evaluate the Efficacy and Safety of KRN321 in Adult Subjects With Low- or Intermediate-1-Risk Myelodysplastic Syndrome
Brief Title: A Clinical Study of KRN321 in Adult Subjects With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRN321-401
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: MDS
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: KRN321

SUMMARY:
This is a multicenter, Randomized, Open-Label, Parallel, Comparative, Dose-Response Study to Evaluate the Efficacy and Safety study of KRN321 of subcutaneous injection in Adult Subjects with Low- or Intermediate-1-Risk Myelodysplastic Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* IPSS low- or intermediate-1-risk MDS diagnosed at enrollment
* Serum EPO concentration ≤ 500 mIU/mL
* Hemoglobin concentration ≤ 9.0 g/dL at the screening examinations

Exclusion Criteria:

* Previous bone marrow or hematopoietic stem cell transplantation
* History of pure red cell aplasia
* Cardiac conditions including angina pectoris, congestive heart failure, uncontrolled arrhythmia and hypertension
* Those who have increased risk of thrombosis during the study
* Uncontrolled diabetes mellitus
* Concurrent active infection or chronic inflammatory disease
* Other causes of anemia
* Previous or concurrent active malignancies other than MDS

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects achieving a erythroid response
Adverse Events as a Measure of Safety

CONTACTS AND LOCATIONS:
Locations (2):
- Saitama, Japan
- Seoul, South Korea